CLINICAL TRIAL: NCT06600919
Title: Effect of Passive Music Therapy Via an App on Anxiety Prevention in ENT Surgery
Acronym: MUSICORL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint-Vincent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSV2024-2
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-09

CONDITIONS: Cervical Surgery; Endonasal Surgery; Otologic Disease; Oropharyngeal Disease; Laryngeal Disease; ENT Surgery; Musical Therapy; Laryngeal Surgery
Keywords: Music therapy; Preoperative anxiety; ENT surgery; Passive music therapy; Randomized controlled trial; Perioperative anxiety; Postoperative pain; Patient care improvement; Clinical research; Music Care® application; Music Care®; Surgical intervention; Anxiety prevention; Music therapy session; Cervical surgery; Endonasal surgery; Otologic surgery; Oropharyngolaryngeal surgery; Musical therapy
MeSH Terms: conditions — Ear Diseases; Laryngeal Diseases; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two parallel arms (intervention group receiving passive music therapy and control group not receiving it)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm: Passive Music Therapy (Experimental): Participants in the Passive Music Therapy arm will receive preoperative music therapy designed to reduce perioperative anxiety. The intervention will involve listening to calming music via headphones for a 20 minutes before entering the operating room.
  Interventions: Other: Preoperative Music Therapy Session
- Control Arm: Standard Care (No Music Therapy) (No Intervention): Participants in the Control Arm will receive standard care without the intervention of passive music therapy.

INTERVENTIONS:
Other: Preoperative Music Therapy Session — Upon admission to the operating room:
  Patients in the music therapy group will undergo a 20-minute music therapy session while lying on a stretcher in a designated room. This session will be conducted using the Music Care® application (https://www.music.care).
  The sessions are standardized and divided into several phases, following a U-shaped sequence. The effect of this U-sequence is first achieved by a phase of reduced tempo, instrumental density, frequency, and sound volume , followed by a phase of reactivation .
  Patients will be allowed to choose the musical style based on their preferences (influenced by their musical tastes and ethnicity). Given the ethnically diverse population of Réunion Island, a wide range of musical preferences is expected.
  Arms: Intervention Arm: Passive Music Therapy

SUMMARY:
Music therapy is a controlled method of listening to music, utilizing its physiological, psychological, and emotional effects on humans during the treatment of illness or trauma. It is considered active when it involves playing musical instruments and passive when it involves listening to music (via headphones, television, stereo systems, etc.).

The benefits of this technique in treating chronic pain (i.e., pain lasting several weeks, such as chronic back pain, osteoarthritis, etc.) have been demonstrated. Numerous studies have also examined the effect of music therapy on acute postoperative pain and anxiety related to surgical interventions. These studies suggest, though without conclusive evidence, that a single session of music therapy just before entering the operating room may reduce postoperative pain and anxiety.

However, all of these studies were limited by relatively small sample sizes (a few hundred patients), leaving some scientific uncertainty regarding the effectiveness of music therapy in the context of surgical interventions.

This research will therefore evaluate the impact of preoperative passive music therapy on perioperative anxiety and postoperative pain, with a larger number of patients included in the study than has been previously reported in the scientific literature.

The primary objective of this study is to assess the impact of preoperative passive music therapy on perioperative anxiety in patients undergoing ENT surgery. MUSICORL is an interventional, randomized study (the assignment to receive or not receive music therapy will be determined by randomization) with two parallel arms. This is a single-center study, conducted at a single French site: Clinique Saint Vincent. A total of 500 subjects will participate in this study. Your participation will last for 2 days; the overall study duration will be 27 months.

To participate in this research, you must be affiliated with a social security system, be over 18 years old, have signed informed consent, and be scheduled for ENT surgery (cervical, endonasal, otologic, oropharyngeal-laryngeal).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older
* Patient has signed informed consent
* Patient scheduled to undergo ENT surgery (cervical, endonasal, otologic, oropharyngeal-laryngeal) at the participating facility
* Patient is affiliated with or a beneficiary of a social security system

Exclusion Criteria:

* Refusal to provide consent
* Patient with severe bilateral hearing loss (> 70 dB HL)
* Patient unable to read, write, or understand French
* Vulnerable patient as defined by Article L1121-6 of the French Public Health Code (CSP)
* Adult patient under guardianship, curatorship, or judicial protection
* Patient unable to personally provide consent as per Article L1121-8 of the CSP or an adult under legal protection
* Pregnant or breastfeeding women as per Article L1121-5 of the CSP
* Patient who has already participated in the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Variation in Anxiety VAS (VAS-A) | From hospital admission to hospital discharge.within an estimated 6 to 24 hours (depending on the average duration of outpatient care)
  Change in the anxiety Visual Analog Scale (VAS-A, ranging from 0 to 10) measured during the hospital stay. The anxiety levels will be recorded at two key time points: admission to the hospital and discharge.

SECONDARY OUTCOMES:
Anxiety VAS (VAS-A) at Key Surgical Phases | Measured at arrival in the operating room and upon exit from the Post-Anesthesia Care Unit (PACU), within an estimated time frame of 2 to 6 hours
  Anxiety levels measured using the Visual Analog Scale (VAS-A, ranging from 0 to 10)
STAI-Y-STATE Anxiety Questionnaire | Measured at hospital admission and hospital discharge, within an estimated time frame of 6 to 24 hours (due to the outpatient nature of the procedure)
  Anxiety levels will be measured using the STAI-Y-STATE questionnaire (State-Trait Anxiety Inventory Form Y), which uses a 4-point Likert scale ranging from 1 to 4 . Higher scores indicate greater levels of anxiety, while lower scores indicate less anxiety. Anxiety scores will be recorded at two key points: upon hospital admission and at discharge.
Total Analgesic Consumption During Hospital Stay | Measured from hospital admission to hospital discharge, within an estimated time frame of 6 to 24 hours (due to the outpatient nature of the procedure).
  The total amount of analgesic medication consumed during the entire hospital stay.
Blood Pressure at Various Time Points | Measured at hospital admission, arrival in the operating room, start of induction, exit from PACU, and hospital discharge, within an estimated time frame of 6 to 24 hours (due to the outpatient nature of the procedure).
  Blood pressure measurements, including both systolic and diastolic values, taken at several critical time points: upon hospital admission, upon arrival in the operating room, at the start of anesthesia induction, upon exit from PACU, and upon hospital discharge.
Surgical and Anesthesia Timeline | During the entire surgical process.
  Key time points during the surgical process will be recorded, including: time of entry into the operating room, start of anesthesia induction, time of incision, time of wound closure, end of anesthesia, exit from the operating room, entry into PACU, and exit from PACU.
Patient and Staff Satisfaction via Likert Scale | Measured at the time of the patient's exit from PACU, within an estimated time frame of 0 to 4 hours after surgery
  Satisfaction levels of both patients and healthcare staff will be evaluated using a 5-point Likert scale (ranging from 1 to 5). Higher scores indicate greater satisfaction, while lower scores indicate less satisfaction.
Medical-Economic Impact | Measured from the start of surgery until hospital discharge, within an estimated time frame of 1 to 6 hours, depending on the specific procedure and recovery time.
  The economic impact will be assessed by measuring the duration of surgery, duration of stay in the PACU, and overall length of hospital stay (measured in minutes).
Variation in Pain VAS (VAS-P) | Measured at hospital admission, arrival in the operating room, exit from PACU, and hospital discharge, within an estimated time frame of 6 to 24 hours (depending on the outpatient procedure).
  Pain levels measured using the Visual Analog Scale (VAS-P, ranging from 0 to 10) at several time points during the hospital stay: upon admission, upon arrival in the operating room, upon exit from the post-anesthesia care unit (PACU), and at hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Vincent, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.music.care/